CLINICAL TRIAL: NCT03421522
Title: Intercostobrachial Nerve Sparing in Breast Cancer Surgery to Reduce Persistent Post-surgical Pain - an International Randomized Controlled Trial
Brief Title: Intercostobrachial Nerve Sparing to Reduce Post-Surgical Pain
Acronym: INSPIRE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: INSPIRE-001
Record Dates: First submitted 2018-01-18; First posted 2018-02-05 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2019-12

CONDITIONS: Post-surgical Pain; Pain, Chronic; Intercostal Pain; Breast Cancer
Keywords: PPSP; ICBN
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: For participants randomized to the ICBN preserving technique, surgeons will perform axillary dissection in which the second ICBN, just inferior to the axillary vein, will be preserved
Who Masked: Participant
Masking Description: Eligible participants will be randomized to one of two treatment groups: 1) ICBN preservation, or 2) usual surgical technique (ICBN sacrifice). Due to the nature of the intervention, it will not be feasible to blind the treating surgeons or the study personnel. The patients, data analysts, and those interpreting the study results will be blinded to treatment allocation.To ensure concealed allocation, eligible patients will be randomized using the randomization function within the REDCap Cloud electronic data capture system. Treatment allocation will be stratified by clinical site to account for systematic differences in surgeons and peri-operative care. To avoid crossover between treatment allocation, randomization will take place in the operating room after the surgeon has confirmed that the participant is a candidate for ICBN preservation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - ICBN preservation (Experimental): For participants randomized to the ICBN preserving technique, surgeons will perform axillary dissection in which the second ICBN, just inferior to the axillary vein, will be preserved.
  Interventions: Other: ICBN preservation surgery
- Control - Usual Care (No Intervention): For participants allocated to the usual surgical care arm, attending surgeons will perform a standard Level 1 and 2 axillary node dissection (sacrifice of the ICBN), either alone or with mastectomy or breast conserving surgery.

INTERVENTIONS:
Other: ICBN preservation surgery — For participants randomized to the ICBN preserving technique, surgeons will perform axillary dissection in which the second ICBN, just inferior to the axillary vein, will be preserved. Surgeons will be asked to indicate whether the ICBN nerve was fully preserved, partially preserved, or sacrificed.
  All study participants will receive anesthetic management at the discretion of the attending physician, which will be documented.
  Arms: Intervention - ICBN preservation

SUMMARY:
Sacrifice of the intercostobrachial nerve (ICBN) during surgery is associated with development of persistent post-surgical pain (PPSP), which affects up to 60% of breast cancer surgery patients. A large, definitive trial is needed to establish whether nerve preservation techniques are effective in reducing post-surgical pain after breast cancer surgery. If the effect of ICBN preservation is consistent with observational studies, the absolute reduction of rates of persistent pain would be considerable.The primary objective is to determine the effect of ICBN preservation, versus usual care, on the prevalence and intensity of PPSP at one year after breast cancer surgery involving axillary lymph node dissection (ALND). Within the larger INSPIRE pilot, we will also be conducting a biomarker sub-study. The objectives of the biomarker sub-study are: 1) to determine the association between pro-inflammatory cytokine levels and the presence and intensity of persistent pain at 3 weeks, and 3 months post-surgery, and) 2) to determine the effect of study intervention on the change in cytokine levels (pre-operative to post-operative) in participants who consent to participate in the sub-study.

DETAILED DESCRIPTION:
A 2016 systematic review that included 30 observational studies (n= 19,813 patients) found high quality evidence that axillary lymph node dissection (ALND) is associated with a 21% absolute risk increase of PPSP (95% CI = 13% to 29%). In many cases of breast cancer, surgery involves axillary approaches; however, preliminary evidence suggests that preservation of the intercostobrachial nerves (ICBN) may reduce the incidence of PPSP after axillary clearance. A 2014 systematic review found 3 small, single-center randomized controlled trials (RCTs), that enrolled a total of 309 patients, and explored the effect of ICBN preservation versus sacrifice during breast cancer surgery. This review found that division of the ICBN was associated with higher risk of sensory deficits, and that nerve preservation techniques increased the median operating time by 5 minutes. Due to limitations of existing evidence, clinical practice guidelines currently provide no recommendations on whether the ICBN should be preserved during axillary lymph node dissection.A large, definitive trial is needed to establish whether nerve preservation techniques are effective in reducing PPSP after breast cancer surgery involving ALND. If all the apparent effect of axillary dissection is associated with lack of ICBN preservation, the absolute reduction of rates of PPSP would be considerable. Furthermore, nerve sparing requires no specialized equipment, suggesting that scalability will be highly feasible.

In addition, there is substantial evidence that neuro-inflammation as a result of neural damage leads to peripheral and central changes that can be described as peripheral and central sensitization, leading to PPSP. As such, we will be conducting a biomarker sub-study as part of the pilot program. Identification of biomarkers to correlate with the development of neuropathic pain may facilitate identification of individuals at risk for development of PPSP at an early stage. The INSPIRE trial provides an important opportunity to compare patients before and after nerve injury to further explore the association of persistent pain with cytokine biomarkers. The findings will improve our mechanistic understanding of PPSP.

ELIGIBILITY:
Pilot Study

Inclusion Criteria:

1. Females aged 18 years and older.
2. Known or suspected invasive breast cancer.
3. Planned ALND (not sentinel lymph node biopsy) either alone or with planned mastectomy or breast conserving surgery.
4. The ICBN is preservable (as confirmed in the OR)
5. Cognitive ability and language skills required to complete the outcome measures.
6. Provision of informed consent.

Exclusion Criteria:

1. The patient has chronic pain or a chronic pain syndrome for which they have received daily medication (i.e. opioid, anti-convulsant, anti-spasmodic, anti-depressant, anti-inflammatory) or routine pain intervention (i.e. nerve blocks) during the past 3 months.

   Note: Chronic pain refers to known chronic pain disorder (i.e. post-herpetic neuralgia, complex regional pain syndrome, fibromyalgia, diabetic neuropathy, post-stroke pain, etc.). The diagnosis for a 'chronic pain syndrome' is outlined by the use of pain medications and interventions. The pain medication must be used by the patient to treat pain. For a pain intervention to be considered routine, it must be given in its prescribed frequency during the past three months (e.g. a patient that has been prescribed to receive a nerve block once a month, received three nerve blocks in the past three months).
2. The patient has a prior history of completing ALND on the ipsilateral side.
3. Detectable metastatic disease at the time of initial diagnosis.
4. Planned bilateral ALND.
5. History of shoulder trauma or pathology on the same side as their breast cancer.
6. Preservation of the ICBN is not possible, in the judgement of the attending surgeon (as confirmed in the OR).
7. Anticipated problems with the patient being available for follow-up.
8. Incarceration.
9. The patient is or may be enrolled in a competing trial.
10. Other reason to exclude the patient, as specified.

Biomarker Sub-Study Eligibility:

All eligible patients who consent to participate in the INSPIRE trial will be asked to participate in the biomarker sub-study. Participants who decline to participate in the biomarker sub-study will still be enrolled into the INSPIRE trial. During the pilot phase of the INSPIRE trial, we will confirm our ability to obtain and analyze blood samples from ≥ 90% of INSPIRE participants.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Persistent post-surgical pain (PPSP) | 12 months
  Post-surgery as defined by the World Health Organization (WHO).
  The WHO's definition requires 4 criteria for the diagnosis of PPSP:
  1. Pain that began after surgery or a tissue trauma is experienced;
  2. The pain is in an area of preceding surgery or tissue trauma,
  3. The pain has persisted for at least three months after surgery, and
  4. The pain is not better explained by an infection, malignancy, a pre-existing pain condition or any other alternative cause.
Moderate-to-severe PPSP | 12 months
  We will establish the severity of PPSP with an item from the Brief Pain Inventory Short Form (BPI-SF), which asks patients to report their 'average' pain intensity rating in the past 24 hrs, on a scale of 0 (no pain) to 10 (maximum pain).
  As per the BPI-SF scoring system, we will define moderate-to-severe pain as scores of ≥4 out of 10.
Biomarker Sub-Study: Cytokine Levels and PPSP | 3 weeks, 3 months
  We will determine the correlation between pro-inflammatory cytokine levels and the presence and intensity of persistent pain at 3 weeks, and 3 months post-surgery
Biomarker Sub-Study: Cytokine Levels Pre and Post-Op | 3 weeks
  We will determine the effect of the study intervention on the change in cytokine levels (pre-operative to post-operative) in participants who consent to participate in the sub-study.

SECONDARY OUTCOMES:
Operative Time | 12 months
  Operative time will be measured from the time of the first incision until the time of closure of the incision.
General physical functioning | 12 months
  Short Form-36 Health Assessment Survey (SF-36) Physical Component Summary score.
  The range of possible scores goes from 0 (worst possible physical functioning) to 100 (best possible physical functioning)
General Mental functioning | 12 months
  Short Form-36 Health Assessment Survey (SF-36) Mental Component Summary score.
  The range of possible scores goes from 0 (worst possible mental functioning) to 100 (best possible mental functioning)
Upper limb-specific physical functioning | 12 months
  The Quick-Disability Arm Shoulder Hand Survey (Quick-DASH).
  An 11-item scale that measures physical function in people with any or multiple musculoskeletal disorders of the upper limb.
  The range of scores goes from 0 (worst possible functioning) to 100 (best possible functioning).
Return to Work | 12 months
  We will document when participants, who were employed before their surgery, return to work.
Adverse Events | 12 months
  All adverse events will be documented on the study specific case report forms. An independent medical monitor will also review each adverse event to determine its relatedness to the surgical treatment.
Pain Interference | 12 months
  Item PAININ18 of the PROMIS will be used to determine the proportion of patients who report somewhat-to-very much pain interference over 12 months post-surgery.
  This item is scored from 0 (not at all) to 4 (very much), and we will use a cut-off value of 2 (somewhat) or higher to define an event.
Use of Prescription Opioids | 12 months
  We will capture the proportion of patients who are prescribed an opioid at 3, 6, 9 and 12-months post-surgery, including the type and dose.
Return to household activities | 12 months
  We will document when participants return to their normal household activities.
Return to leisure activities | 12 months
  We will document when participants return to their normal leisure activities.
Return to pre-surgical functioning | 12 months
  We will document when participants achieve 80% of their pre-surgery function, as measured on a percentage scale of 0% (no function) to 100% (full pre-surgical function).

CONTACTS AND LOCATIONS:
Overall Officials: Susan Dr Reid, Principal Investigator — Hamilton Health Sciences - Juravinski Hospital; Jason Busse, Principal Investigator — McMaster Michael DeGroote Centre for National Pain Research and Care; Sheila Sprague, Principal Investigator — McMaster
Locations (1):
- Juravinski Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersen KG, Kehlet H. Persistent pain after breast cancer treatment: a critical review of risk factors and strategies for prevention. J Pain. 2011 Jul;12(7):725-46. doi: 10.1016/j.jpain.2010.12.005. Epub 2011 Mar 24. PMID 21435953
- [Background] Gureje O, Von Korff M, Simon GE, Gater R. Persistent pain and well-being: a World Health Organization Study in Primary Care. JAMA. 1998 Jul 8;280(2):147-51. doi: 10.1001/jama.280.2.147. PMID 9669787
- [Background] Wang L, Guyatt GH, Kennedy SA, Romerosa B, Kwon HY, Kaushal A, Chang Y, Craigie S, de Almeida CPB, Couban RJ, Parascandalo SR, Izhar Z, Reid S, Khan JS, McGillion M, Busse JW. Predictors of persistent pain after breast cancer surgery: a systematic review and meta-analysis of observational studies. CMAJ. 2016 Oct 4;188(14):E352-E361. doi: 10.1503/cmaj.151276. Epub 2016 Jul 11. PMID 27402075
- [Background] Warrier S, Hwang S, Koh CE, Shepherd H, Mak C, Carmalt H, Solomon M. Preservation or division of the intercostobrachial nerve in axillary dissection for breast cancer: meta-analysis of randomised controlled trials. Breast. 2014 Aug;23(4):310-6. doi: 10.1016/j.breast.2014.01.014. Epub 2014 Feb 24. PMID 24582033
- [Background] Gherghe M, Bordea C, Blidaru A. Sentinel lymph node biopsy (SLNB) vs. axillary lymph node dissection (ALND) in the current surgical treatment of early stage breast cancer. J Med Life. 2015 Apr-Jun;8(2):176-80. PMID 25866575
- [Background] Treede RD, Rief W, Barke A, Aziz Q, Bennett MI, Benoliel R, Cohen M, Evers S, Finnerup NB, First MB, Giamberardino MA, Kaasa S, Kosek E, Lavand'homme P, Nicholas M, Perrot S, Scholz J, Schug S, Smith BH, Svensson P, Vlaeyen JWS, Wang SJ. A classification of chronic pain for ICD-11. Pain. 2015 Jun;156(6):1003-1007. doi: 10.1097/j.pain.0000000000000160. No abstract available. PMID 25844555
- [Background] Tan G, Jensen MP, Thornby JI, Shanti BF. Validation of the Brief Pain Inventory for chronic nonmalignant pain. J Pain. 2004 Mar;5(2):133-7. doi: 10.1016/j.jpain.2003.12.005. PMID 15042521
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Angst F, Aeschlimann A, Stucki G. Smallest detectable and minimal clinically important differences of rehabilitation intervention with their implications for required sample sizes using WOMAC and SF-36 quality of life measurement instruments in patients with osteoarthritis of the lower extremities. Arthritis Rheum. 2001 Aug;45(4):384-91. doi: 10.1002/1529-0131(200108)45:43.0.CO;2-0. PMID 11501727
- [Background] Jenkinson C, Stewart-Brown S, Petersen S, Paice C. Assessment of the SF-36 version 2 in the United Kingdom. J Epidemiol Community Health. 1999 Jan;53(1):46-50. doi: 10.1136/jech.53.1.46. PMID 10326053
- [Background] Busse JW, Bhandari M, Guyatt GH, Heels-Ansdell D, Mandel S, Sanders D, Schemitsch E, Swiontkowski M, Tornetta P 3rd, Wai E, Walter SD; SPRINT Investigators. Use of both Short Musculoskeletal Function Assessment questionnaire and Short Form-36 among tibial-fracture patients was redundant. J Clin Epidemiol. 2009 Nov;62(11):1210-7. doi: 10.1016/j.jclinepi.2009.01.014. Epub 2009 Apr 11. PMID 19364637
- [Background] Mintken PE, Glynn P, Cleland JA. Psychometric properties of the shortened disabilities of the Arm, Shoulder, and Hand Questionnaire (QuickDASH) and Numeric Pain Rating Scale in patients with shoulder pain. J Shoulder Elbow Surg. 2009 Nov-Dec;18(6):920-6. doi: 10.1016/j.jse.2008.12.015. Epub 2009 Mar 17. PMID 19297202
- [Background] Trudel JG, Rivard M, Dobkin PL, Leclerc JM, Robaey P. Psychometric properties of the Health Utilities Index Mark 2 system in paediatric oncology patients. Qual Life Res. 1998 Jul;7(5):421-32. doi: 10.1023/a:1008857920624. PMID 9691722
- [Background] Brodke DJ, Saltzman CL, Brodke DS. PROMIS for Orthopaedic Outcomes Measurement. J Am Acad Orthop Surg. 2016 Nov;24(11):744-749. doi: 10.5435/JAAOS-D-15-00404. PMID 27661391
- [Background] Fries JF, Bruce B, Cella D. The promise of PROMIS: using item response theory to improve assessment of patient-reported outcomes. Clin Exp Rheumatol. 2005 Sep-Oct;23(5 Suppl 39):S53-7. PMID 16273785
- [Background] Khan JS, Devereaux PJ, LeManach Y, Busse JW. Patient coping and expectations about recovery predict the development of chronic post-surgical pain after traumatic tibial fracture repair. Br J Anaesth. 2016 Sep;117(3):365-70. doi: 10.1093/bja/aew225. PMID 27543531
- [Background] Reininga IH, Brouwer S, Dijkstra A, Busse JW, Ebrahim S, Wendt KW, El Moumni M. Measuring illness beliefs in patients with lower extremity injuries: reliability and validity of the Dutch version of the Somatic Pre-Occupation and Coping questionnaire (SPOC-NL). Injury. 2015 Feb;46(2):308-14. doi: 10.1016/j.injury.2014.08.042. Epub 2014 Sep 16. PMID 25441575
- [Background] Busse JW, Bhandari M, Guyatt GH, Heels-Ansdell D, Kulkarni AV, Mandel S, Sanders D, Schemitsch E, Swiontkowski M, Tornetta P 3rd, Wai E, Walter SD; SPRINT Investigators & the Medically Unexplained Syndromes Study Group. Development and validation of an instrument to predict functional recovery in tibial fracture patients: the Somatic Pre-Occupation and Coping (SPOC) questionnaire. J Orthop Trauma. 2012 Jun;26(6):370-8. doi: 10.1097/BOT.0b013e31822421e2. PMID 22011635
- [Background] Abdullah TI, Iddon J, Barr L, Baildam AD, Bundred NJ. Prospective randomized controlled trial of preservation of the intercostobrachial nerve during axillary node clearance for breast cancer. Br J Surg. 1998 Oct;85(10):1443-5. doi: 10.1046/j.1365-2168.1998.00843.x. PMID 9782034
- [Background] Salmon RJ, Ansquer Y, Asselain B. Preservation versus section of intercostal-brachial nerve (IBN) in axillary dissection for breast cancer--a prospective randomized trial. Eur J Surg Oncol. 1998 Jun;24(3):158-61. doi: 10.1016/s0748-7983(98)92793-7. PMID 9630850
- [Background] Torresan RZ, Cabello C, Conde DM, Brenelli HB. Impact of the preservation of the intercostobrachial nerve in axillary lymphadenectomy due to breast cancer. Breast J. 2003 Sep-Oct;9(5):389-92. doi: 10.1046/j.1524-4741.2003.09505.x. PMID 12968959
- [Background] Sprague S, Leece P, Bhandari M, Tornetta P 3rd, Schemitsch E, Swiontkowski MF; S.P.R.I.N.T. Investigators. Limiting loss to follow-up in a multicenter randomized trial in orthopedic surgery. Control Clin Trials. 2003 Dec;24(6):719-25. doi: 10.1016/j.cct.2003.08.012. PMID 14662277
- [Background] Madden K, Scott T, McKay P, Petrisor BA, Jeray KJ, Tanner SL, Bhandari M, Sprague S. Predicting and Preventing Loss to Follow-up of Adult Trauma Patients in Randomized Controlled Trials: An Example from the FLOW Trial. J Bone Joint Surg Am. 2017 Jul 5;99(13):1086-1092. doi: 10.2106/JBJS.16.00900. PMID 28678121
- [Background] Zhang Y, Alyass A, Vanniyasingam T, Sadeghirad B, Florez ID, Pichika SC, Kennedy SA, Abdulkarimova U, Zhang Y, Iljon T, Morgano GP, Colunga Lozano LE, Aloweni FAB, Lopes LC, Yepes-Nunez JJ, Fei Y, Wang L, Kahale LA, Meyre D, Akl EA, Thabane L, Guyatt GH. A systematic survey of the methods literature on the reporting quality and optimal methods of handling participants with missing outcome data for continuous outcomes in randomized controlled trials. J Clin Epidemiol. 2017 Aug;88:67-80. doi: 10.1016/j.jclinepi.2017.05.016. Epub 2017 Jun 1. PMID 28579378
- See also: Canadian Cancer Statistics — http://www.cancer.ca
- See also: Visnjevac OM, B. Postmastectomy pain syndrome: an unrecognized annual billion dollar national financial burden. J Pain 2013;14 — http://dx.doi.org/10.1016/j.jpain.2013.01.487
- See also: K. M. Intercostobrachial syndrome after nerve-sparing axillary lymph node dissection. Eur J Cancer. 2014;50:S127. — https://www.ncbi.nlm.nih.gov/pubmed/25307709
- See also: Busse JW, Bhandari M, Einhorn TA, Schemitsch E, Heckman JD, Tornetta P, 3rd, et al. Re-evaluation of low intensity pulsed ultrasound in treatment of tibial fractures (TRUST): randomized clinical trial. Bmj. 2016;355:i5351. — http://www.bmj.com/content/355/bmj.i5351
- See also: Hamner J, Dewitt B. The Development of a Preference-based Scoring System for PROMIS (PROPr): A Technical Report v 1.1. [Internet] 2017;available from: http://janelhanmer.pitt.edu/documents/technicalreportv1.1.pdf (accessed August 29, 2017). — http://janelhanmer.pitt.edu/ProPr.html